CLINICAL TRIAL: NCT00147355
Title: An Open-label, Randomised Study Comparing the Uptake of rIL-2 in HIV-1 Infected Individuals Receiving Different Combinations of Antiemetics and Analgesic Agents During rIL-2 Dosing in ESPRIT: Toxicity Substudy of ESPRIT: TOXIL-2 Substudy
Brief Title: Toxicity Substudy of Evaluation of Subcutaneous Proleukin in a Randomised International Trial (ESPRIT): TOXIL-2 Substudy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 28 of 168 patients only were enrolled, numbers too low to be conclusive
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ESPRIT TOXIL-2 UNSW PSO 6361; ACTR012605000407695
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: rIL-2-toxicity; interleukin-2 therapy; HIV; Toxicity substudy of ESPRIT
MeSH Terms: conditions — HIV Infections | interventions — Ondansetron; Ibuprofen; Acetaminophen; Metoclopramide; Codeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Other): Ondansetron 4mg bid + Ibuprofen 200mg qds + paracetamol 1g qds days 1-6 inclusive of rIL-2 dosing cycle
  Interventions: Drug: ondansetron, ibuprofen, paracetamol
- B (Other): Ondansetron 4mg bid + codeine phosphate 15mg tds + Ibuprofen 200mg qds + paracetamol 1g qds days 1-6 inclusive of rIL-2 dosing cycle
  Interventions: Drug: Ondansetron, ibuprofen, paracetamol
- D (Other): metoclopramide 10mg qds + codeine phosphate 15mg tds + Ibuprofen 200mg qds + paracetamol 1g qds days 1-6 inclusive of rIL-2 dosing cycle
  Interventions: Drug: Metoclopramide, codeine phosphate, ibuprofen, paracetamol
- C (Other): metoclopramide 10mg qds + Ibuprofen 200mg qds + paracetamol 1g qds days 1-6 inclusive of rIL-2 dosing cycle
  Interventions: Drug: metoclopramide, ibuprofen, paracetamol

INTERVENTIONS:
Drug: ondansetron, ibuprofen, paracetamol — ondansetron 4mg bid + Ibuprofen 200mg qds + paracetamol 1g qds days 1-6 inclusive of rIL-2 dosing cycle
  Arms: A
Drug: Ondansetron, ibuprofen, paracetamol — Ondansetron 4mg bid + codeine phosphate 15mg tds + Ibuprofen 200mg qds + paracetamol 1g qds days 1-6 inclusive of rIL-2 dosing cycle
  Arms: B
Drug: metoclopramide, ibuprofen, paracetamol — metoclopramide 10mg qds + Ibuprofen 200mg qds + paracetamol 1g qds days 1-6 inclusive of rIL-2 dosing cycle
  Arms: C
Drug: Metoclopramide, codeine phosphate, ibuprofen, paracetamol — metoclopramide 10mg qds + codeine phosphate 15mg tds + Ibuprofen 200mg qds + paracetamol 1g qds days 1-6 inclusive of rIL-2 dosing cycle
  Arms: D

SUMMARY:
This substudy is an open-label, randomised study comparing the uptake of recombinant interleukin-2 (rIL-2) in HIV-1 infected individuals receiving different combinations of antiemetics and analgesic agents during rIL-2 dosing in ESPRIT. The design is a factorial one with 4 arms. All patients will receive regular ibuprofen and paracetamol from days 1-6 of the rIL-2 dosing cycle; in addition, patients will be randomised to receive one of two antiemetic combinations, i.e. ondansetron or metoclopramide with or without low dose codeine phosphate as an additional analgesic agent.

DETAILED DESCRIPTION:
The research is a randomised open-label substudy of ESPRIT. The substudy is exploring whether the amount of rIL-2 taken during a dosing cycle of rIL-2 can be increased through controlling the predictable side-effects of rIL-2 better. This is a four arm study with a factorial design; patients will be randomised to one of four arms. Each arm consists of different combinations of adjunctive agents. Each patient will receive paracetamol and ibuprofen prophylactically throughout the cycle, the other adjunctive agents prescribed will vary according to which arm the patient is randomised to, but the antiemetic used will be either ondansetron or metoclopramide with or without low dose codeine phosphate as an additional analgesic agent. The primary end-point is the percentage of planned rIL-2 actually taken during the cycle. Secondary end-points include safety, side-effects of rIL-2 and the adjunctive agents, CD4+ T-cell changes and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

Patients participating in ESPRIT and randomised to the rIL-2 arm, who:

1. Are not at CD4+ T-cell target for the protocol
2. Have not received rIL-2 for > 2 months
3. Have reported both GI upset and constitutional side-effects as one of the reasons for either dose modifying in prior cycles or unwillingness to receive further rIL-2
4. Are considered by the Investigator as medically safe to receive further dosing with rIL-2
5. Are willing to receive further dosing with rIL-2 at the dose specified by the Investigator
6. Are willing to sign informed consent to participate in the substudy

Exclusion Criteria:

1. All exclusions for the receipt of rIL-2 on ESPRIT
2. Known allergy to non-steroidal anti-inflammatory drugs (NSAIDs), opiates, 5HT-3 (serotonin-3) inhibitors, anti-dopaminergic antiemetics, or any other components of the proposed adjunct regimens.
3. Use of other NSAIDs (cyclooxygenase-2 [COX-2] inhibitors, corticosteroids) or opiate analgesics within two weeks of rIL-2 dosing. Use of low dose aspirin as a cardio-protective agent is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-11; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
percentage of planned rIL-2 taken during the first rIL-2 dosing cycle while participating in this substudy. | 6 months
  we are comparing the percentage of planned rIL-2 taken when randomised to one of the four combinations used as adjunctive therapies to alleviate the known side-effects of rIL-2

SECONDARY OUTCOMES:
Patterns of rIL-2 cycling frequency in the six months after randomisation into the substudy | 6 months
  to explore the patterns of rIL-2 and see if the different adjuntive regimens increase tolerability such that more rIL-2 is taken
Percentage of planned rIL-2 taken during the cycles after the first cycle | 6 mths
  this is to assess whether the adjuncts to which the patient was randomised as part of this substudy impact on better tolerability of cycles of rIL-2 beyond the first
Mean difference in rIL-2 taken during each cycle in the six-month period following randomisation into this substudy and rIL-2 uptake during the last dosing cycle immediately prior to participation in the substudy | 6 months
  to see if the adjuncts to which the patient is randomised improve amount of rIL-2 taken compared to the cycle taken prior to enrollment in this substudy
Number of patients with dose modifications during the cycle due to toxicity | 6 months
  to assess whether the adjuncts to which they were randomised reduced the amount of rIL-2 dose modification during the rIL-2 cycle
Number of patients with grade 1-4 constitutional upset (defined as any or all of the following: flu-like illness/fever/myalgia/arthralgia/headache) and/or GI upset and/or evidence of capillary leak syndromes | 6 months
  to assess the impact of the randomised adjuntive agents on the predictable side-effects of rIL-2
Grade 1-4 creatinine and sodium changes during and after rIL-2 dosing; | 6 months
  to assess the impact of the randomised adjuntive agents on the predictable effects of rIL-2 in regards to salt and water homeostasis and renal function
Changes in quality of life during and after rIL-2 | 6 months
  to assess whether the use of different adjunctive agents impacted on the tolerability of rIL-2 during the cycle and post as perceived by the patients qOL
Incidence of SAE and AE | 6 months
  to assess the incidence of SAE and AEs that are rIL-2 (captured for the main study) and adjunctive agents

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Pett, M.D, Principal Investigator — Kirby Institute, Faculty of Medicine, University of New South Wales, Sydney, Australia
Locations (16):
- Argentina (8):
  - Hospital General de Agudos JM Ramos Mejia, Buenos Aires, Buenos Aires
  - FUNCEI, Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires
  - Hospital Prof. Alejandro Posadas, Buenos Aires
  - Hospital Interzonal de Agudos San Juan de Dios, La Plata
  - Hospital Interzonal General de Agudos Oscar Alende, Mar del Plata
  - Hospital Central, Mendoza
  - CAICI, Rosario
- Australia (7):
  - St. Vincent's Hospital, Sydney, New South Wales
  - AIDS Medical Unit, Brisbane, Queensland
  - Cairns Base Hospital, Cairns, Queensland
  - Gold Coast Sexual Health Clinic, Gold Coast, Queensland
  - Nambour Hospital, Nambour, Queensland
  - Carlton Clinic, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Kaplan Medical Center, Rehovot, Israel

REFERENCES:
- See also: National Centre in HIV Epidemiology and Clinical Research Homepage — http://www.med.unsw.edu.au/nchecr/